CLINICAL TRIAL: NCT02183103
Title: Influence of a High Fat Breakfast in the Pharmacokinetics of UH-AC62MU (Rapid Release Tablet) Given as an Oral Single Dose of 7.5 mg in Healthy Subjects (Two Way, Crossover, Randomized, Open)
Brief Title: Influence of a High Fat Breakfast in the Pharmacokinetics of UH-AC62MU in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.224
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- meloxicam rapid release tablet after an overnight fast (Active Comparator)
  Interventions: Drug: meloxicam rapid release tablet, 12mg, UH AC62MU
- meloxicam rapid release tablet after high fat breakfast (Experimental)
  Interventions: Drug: meloxicam rapid release tablet, 12mg, UH AC62MU

INTERVENTIONS:
Drug: meloxicam rapid release tablet, 12mg, UH AC62MU

SUMMARY:
Influence of a high fat breakfast in the pharmacokinetic profile of the 7.5 mg meloxicam rapid releases tablet

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Written informed consent according good clinical practice (GCP) and local legislation
* Age >=18 and <=50 years
* Broca >= -20% and <= +20%

Exclusion Criteria:

* Any finding of the medical examination (blood pressure, pulse rate and electrocardiogram (ECG)) deviating from the normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorder
* Surgery of gastro-intestinal tract (except appendectomy)
* Disease of central nervous system (such as epilepsy) or psychiatric disorders or neurological disorder
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life ( >24h) (<=1month prior to administration)
* Use of any drugs which might influence the results of the trial (<=10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 2 months prior to administration or during the trial)
* Smokers ( >10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (>60g/day)
* Drug abuse
* Blood donation (<= 1 month prior to administration or during the trial)
* Excessive physical activities (<= 5 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* History of hemorrhagic diatheses
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma

For female:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. sterilization, intrauterine device (IUD), oral contraceptives
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 1999-04; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | predose and up to 96 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from time zero to infinity (AUC 0-infinity) | predose and up to 96 hours after drug administration

SECONDARY OUTCOMES:
Time to achieve Cmax (tmax) | predose and up to 96 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from time zero to t (AUC 0-t) | predose and up to 96 hours after drug administration
Terminal rate constant in plasma (λz) | predose and up to 96 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | predose and up to 96 hours after drug administration
Mean residence time of the analyte total (MRT tot) | predose and up to 96 hours after drug administration
Apparent clearance of the analyte in plasma following extravascular administration (CL/F) | predose and up to 96 hours after drug administration
Apparent volume of distribution during the terminal phase λz following extravascular administration (Vz/F) | predose and up to 96 hours after drug administration
Number of patients with abnormal changes in laboratory values | Baseline, 96 hours after drug administration
Number of Participants with Adverse Events | Up to day 5 after last drug administration
Number of patients with abnormal changes from baseline in ECG | Baseline, day 5 after last drug administration
Number of patients with abnormal changes from baseline in physical examination | Baseline, day 5 after last drug administration